CLINICAL TRIAL: NCT05163756
Title: A Multi-center, Double-blind, Randomized, Parallel, Active-controlled, Non-inferiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW1903 in Patients With Gastritis
Brief Title: To Evaluate the Efficacy and Safety of DW1903 in Acute and Chronic Gastritis Patient
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1903-301
Record Dates: First submitted 2021-12-07; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Gastritis Acute; Gastritis Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DW1903(Test) (Experimental): once a day, q.d. PO / DW1903 + Placebo of DW1903-R1
  Interventions: Drug: DW1903
- DW1903-R1(Reference) (Active Comparator): once a day, q.d. PO / Placebo of DW1903 + DW1903-R1
  Interventions: Drug: DW1903-R1

INTERVENTIONS:
Drug: DW1903 — q.d. PO, DW1903 + Placebo of DW1903-R1
  Arms: DW1903(Test)
Drug: DW1903-R1 — q.d. PO, Placebo of DW1903 + DW1903-R1
  Arms: DW1903-R1(Reference)

SUMMARY:
A Multi-center, Double-blind, Randomized, Parallel, Active-controlled, Non-inferiority, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DW1903 in Patients with Gastritis

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with acute or chronic gastritis in a gastroscopy performed within 7 days prior to administration of this trial.
* At least one or more erosions have been identified on gastroscopy.
* Patients who decided to voluntarily participate in this trial and agreed in writing.

Exclusion Criteria:

* Patients who can not undergo gastroscopy
* Peptic ulcer (except scarring) and reflux esophagitis
* Patients who have had gastric acid suppression surgery or stomach/esophagus surgery (except for simple perforation surgery and appendectomy)
* Patients with a history of gastrointestinal malignancies
* Zollinger-Ellison syndrome patients
* Patient with spontaneous coagulation disorder
* Patients with an allergic or hypersensitive response to a study drug
* Patients with a potential pregnancy.
* Patients who had clinically significant abnormalities in the screening test.
* Pregnant and lactating women
* Those currently taking other study drugs
* patients who were judged to be ineligible for the trial by the principle investigator and the person in charge.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
The efficacy rate on gastroscopy | Week 0, Week2
  The efficacy rate is obtained from the following formula using the subject whose erroneous score is improved by 50% or more as compared with before the study drug administration.
  The efficacy rate(%) = (number of effective cases)/(all cases) x 100
  Effective case is determined by the grade change of erosion. A case in which the grade changes from 4 to 2 or 1, from 3 to 1, or from 2 to 1 is judged as an effective case.

SECONDARY OUTCOMES:
Cure rate on gastroscopy | Week 0, Week2
  Judging from the gastroscopic examination as normal (no erosion), the cure rate is obtained as follows.
  Cure rate(%) = (number of cures(no erosion))/(all cases) x 100

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Ansan Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan for IPD.

REFERENCES:
- [Derived] Kim JH, Jung HY, Yoo IK, Park SY, Kim JG, Sung JK, Jang JS, Cheon GJ, Kim KO, Kim TO, Lee ST, Cho KB, Chun HJ, Park JJ, Park MI, Jang JY, Jeon SW, Cho JW, Kang DH, Kim GH, Kim JJ, Kim SG, Kim N, Lee YC, Hong SJ, Kim HS, Lee S, Lee SW. Evaluation of the Efficacy and Safety of DW1903 in Patients with Gastritis: A Randomized, Double-Blind, Noninferiority, Multicenter, Phase 3 study. Gut Liver. 2024 Jan 15;18(1):70-76. doi: 10.5009/gnl220446. Epub 2023 Jun 13. PMID 37309193